CLINICAL TRIAL: NCT07251348
Title: The Effect of Progressive Relaxation and Psychoeducation on Perceived Stress and Hope in Patients With Hematologic Malignancies: A Non-Randomized Study
Brief Title: Progressive Relaxation and Psychoeducation in Patients With Hematological Malignancies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Tuba KORKMAZ ASLAN, ASSOCIATE PROFESSOR, Necmettin Erbakan University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: NEÜ-SBF-TKA-02
Record Dates: First submitted 2025-09-11; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hematological Cancer
Keywords: hematologic malignancy; progressive relaxation; psychoeducation; stress; hope
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Muscle Relaxation; Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Progressive relaxation group; n=25: After the pre-test, 6 sessions (2 sessions per week) were planned for 3 weeks for individuals in this group. Each session will be conducted individually with patients, face-to-face, and will last 40-45 minutes. The post-test was administered after 3 weeks.
  psychoeducation group; n=25: After the pre-test, 6 sessions (2 sessions per week) were planned for 3 weeks for the individuals in this group. Each session will be conducted individually with patients, face-to-face, and will last 40-45 minutes. A post-test was administered after 3 weeks. Four expert opinions were obtained regarding the content.
  routine nursing care group: no intervention n=25: The 'Perceived Stress Level' scale and the 'Herth Hope Index' scale will be administered after the initial interview.
  Routine nursing care was provided.After 3 weeks, the 'Perceived Stress Level' scale and the 'Herth Hope Index' scale will be administered after the
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Progressive relaxation (Active Comparator): Progressive relaxation; n=25: After the pre-test, 6 sessions (2 sessions per week) were planned for 3 weeks for individuals in this group. Each session will be conducted individually with patients, face-to-face, and will last 40-45 minutes. The post-test was administered after 3 weeks.
  PROGRESSIVE RELAXATION SESSION TITLES:
  1. SESSION: Introduction, Establishing Trust and the Concept of Relaxation
  2. SESSION: Coping with a Cancer Diagnosis & Introduction to the Progressive Relaxation Technique
  3. SESSION: Progressive Muscle Relaxation Application - Upper Body3
  4. SESSION: Progressive Muscle Relaxation - Lower Body
  5. SESSION: Whole Body Relaxation - Reinforcing the Application
  6. SESSION: Integrating Progressive Relaxation into Daily Life & Closing
  Interventions: Behavioral: Muscle Relaxation
- psychoeducation (Active Comparator): psychoeducation; n=25: After the pre-test, 6 sessions (2 sessions per week) were planned for 3 weeks for the individuals in this group. Each session will be conducted individually with patients, face-to-face, and will last 40-45 minutes. A post-test was administered after 3 weeks. Four expert opinions were obtained regarding the content.
  PSYCHOEDUCATION SESSION TITLES:
  1. SESSION: INTRODUCTION AND PROGRAM OVERVIEW 2nd SESSION: UNDERSTANDING THE DISEASE - EMPOWERING THROUGH KNOWLEDGE 3rd SESSION: IDENTIFYING PERCEIVED STRESS AND ITS EFFECTS 4. SESSION: COPING WITH STRESS AND INTRODUCTION TO HOPE 5. SESSION: UNDERSTANDING AND STRENGTHENING HOPE 6. SESSION: INTERNALIZING WHAT HAS BEEN LEARNED, MAINTAINING AND EVALUATING
  Interventions: Behavioral: psychoeducation or Atomoxetine or stimulants according to ADHD severity
- routine nursing care (No Intervention): routine nursig care; n=25 No intervention was performed after the pre-test; routine nursing care was administered. The post-test was administered after 3 weeks.

INTERVENTIONS:
Behavioral: Muscle Relaxation — Progressive relaxation is a relaxation technique based on tensing and relaxing muscles in sequence. The goal is to achieve physical and mental relaxation by feeling the difference between tension and relaxation. It is frequently used for stress, anxiety, sleep problems, and psychosomatic disorders. When practiced regularly, it increases a person's ability to relax and contributes to their overall well-being.
  * Teaching progressive relaxation exercises to individuals diagnosed with cancer and supporting psychological well-being by reducing stress levels and increasing hope levels through these exercises (emotional gain)
  * Reducing muscle tension and providing physical relaxation (psychomotor gain)
  * To reduce stress and anxiety (emotional gain)
  * To increase body awareness (emotional gain)
  * To teach mental and physical relaxation (psychomotor gain)
  * To provide emotional relief (emotional gain)
  * To develop self-relaxation skills (psychomotor gain)
  Arms: Progressive relaxation
Behavioral: psychoeducation or Atomoxetine or stimulants according to ADHD severity — Psychoeducation is a structured educational process that provides individuals with information about mental illnesses, ways to cope with stress, and healthy living skills. The goal is to help the person understand their illness and symptoms, learn coping methods, and increase their compliance with treatment. It has both an informative and a supportive aspect.
  INTERVENTION B (PSYCHOEDUCATION) GROUP APPLICATION:
  * A total of 6 sessions will be held with patients in intervention group B, twice a week for 3 weeks.
  * Each session will last an average of 45 minutes.
  * The 'Perceived Stress Level' scale and the 'Herth Hope Index' scale will be administered after the first session.
  * The 'Perceived Stress Level' scale and the 'Herth Hope Index' scale will be administered after the final session.
  Arms: psychoeducation

SUMMARY:
This study will be conducted to determine the effect of progressive relaxation and psychoeducation on perceived stress and hope in patients with hematological malignancies

DETAILED DESCRIPTION:
Being healthy requires being in a state of complete physical and mental well-being. Therefore, mental and physical well-being must be maintained together. While each individual already has different stressors, the fact that hematological malignancies are chronic and immune-mediated diseases increases the stress factors perceived by individuals, and the difficulty and uncertainty of the process reduces their level of hope. This triggers the use of ineffective coping methods. Patients with high perceived stress levels and declining hope levels are unable to adequately manage the disease process. Consequently, mortality and morbidity rates increase. This experimentally planned study will be conducted between February 2026 and November 2026 at the Adult Inpatient Hematology Clinic of Gazi University Faculty of Medicine Hospital. The study will involve 75 individuals hospitalized at the clinic who meet the inclusion criteria. It is a non-randomized study with 2 intervention groups and 1 control group. Intervention group A (progressive relaxation group, n=25), intervention group B (psychoeducation, n=25), and control group (routine care, n=25). Patients in intervention group A will undergo a 3-week, 6-session progressive relaxation exercise program, conducted individually and face-to-face. Intervention Group B will receive a 3-week, 6-session, individual, face-to-face psychoeducation program. The control group will receive 3 weeks of routine nursing care identical to that provided to the other groups. In this study, which will include pre- and post-tests, data will be collected face-to-face using the perceived stress level scale and the Herth hope index scale. The primary objective of this study is to examine the effects of progressive relaxation and psychoeducation interventions on perceived stress and hope levels in patients with hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Diagnosis of hematologic malignancy
3. Ability to read and write
4. Volunteer to participate in the study

Exclusion Criteria:

1. Dementia and/or organic mental disorder
2. Sensory loss related to vision and hearing
3. Communication barrier
4. Physical disability
5. Respiratory distress
6. Bone marrow transplant procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Herth hope index level scale | 9 months
  Herth Hope Index: Developed by Kaye Herth (1992), its validity and reliability in Turkish were studied by Aslan and colleagues (2007). The scale consists of a total of 12 items: "Future" (questions 1, 2, 6, 11), "Positive readiness and expectation" (questions 4, 7, 10, 12), and "Connections with oneself and others" (questions 3, 5, 8, 9).
perceived stress level scales | 9 months
  PERCEIVED STRESS SCALE: The adaptation of the perceived stress scale developed by Cohen, Kamarck, and Mermelsten (1983) into Turkish was carried out by Eskin et al. (2013). The perceived stress scale, consisting of a total of 14 items, aims to measure how stressful individuals perceive their life situations to be..

IPD SHARING:
Plan to Share IPD: No